CLINICAL TRIAL: NCT01152333
Title: The Role of GLP-1 in Satiety Perception in Humans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is delayed. It was not funded.
Sponsor: University of Washington (Other)
Collaborators: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Ellen Schur, MD, MS, Ellen A Schur, MD, MS, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 37919-D; 1R03DK083502-01A1 (NIH)
Record Dates: First submitted 2010-06-15; First posted 2010-06-29 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Appetite Regulation; Obesity
MeSH Terms: conditions — Obesity | interventions — exendin (9-39); Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exendin (9-39) Acetate (Active Comparator): Exendin (9-39) is a synthetic peptide that acts as an antagonist to the GLP-1 receptor. Exendin (9-39) will be diluted in saline 0.9% and administered through IV infusion once for a maximum of 2.5 hours in length at 600-750 pM/kg/min.
  Interventions: Drug: Exendin-(9-39) Acetate
- Saline (Placebo Comparator): Saline 0.9% will be used as the control infusion.
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Exendin-(9-39) Acetate — Exendin (9-39) will be diluted in saline 0.9% and administered through IV infusion once for a maximum of 2.5 hours in length.
  Arms: Exendin (9-39) Acetate
Drug: Saline 0.9% — Saline will be administered through IV infusion once for a maximum of 2.5 hours in length
  Other Names: Sodium chloride (NaCl)
  Arms: Saline

SUMMARY:
Scientists have discovered a number of hormones that control our feelings of hunger and fullness. One particular hormone, called GLP-1, has been associated with feelings of hunger and fullness. The overall purpose of this study is to look more closely at how GLP-1 changes these feelings and to observe how these hormones affect the brain's function. To do this, volunteers will be asked to come to the clinic for a screening visit, and 2 study visits. This is an outpatient study with a screening visit which will last about an hour and the two subsequent study visits for about 3 hours each. During the study, patients will receive a drug that blocks the effect of a hormone made in the gut. We will take a series of blood samples to measure hormones and use functional magnetic resonance imaging (MRI) to take pictures of the brain. Understanding the action of these hormones in the brain may eventually lead to new ways to help people avoid obesity or lose weight.

DETAILED DESCRIPTION:
Many times each day, we see food or representations of food and evaluate whether or not the food looks good to us. If it does, we then balance external factors, such as the social situation or time of day, against internal signals about our hunger state in order to decide what and when to eat. However, recent functional magnetic resonance imaging (fMRI) studies suggest that internal signals, such as hormones regulating appetite and satiety, govern our food intake in part by acting on neural circuits to affect whether a given food appears appetizing at that moment. In addition, photographs of food perceived to be "fattening" activate brain regions involved in appetite and reward processing, including the hypothalamus, nucleus accumbens, and orbital frontal cortex. This activity is potently reduced by food intake, suggesting that it reflects underlying brain mechanisms involved in satiety. We now propose to study the mechanism of these changes in brain activity by asking if they are directly related to the action of glucagon-like peptide-1 (GLP-1), a satiety signal. GLP-1 is released by cells in the gut in response to nutrients, suppressing food intake, and its actions can be blocked by a GLP-1 receptor antagonist, exendin-[9-39]. In 2 randomized, controlled, crossover studies, we will assess whether exendin-[9-39] infusions reverse GLP-1-mediated effects on food intake and on brain response to visual food cues. Our scientific aims are to 1) observe the effect of exendin (9-39) on blocking GLP-1-mediated satiety in humans and assess its effect on food intake in humans for the first time (to our knowledge) and 2) to test whether endogenous GLP-1 signaling is required for the effect of a meal to reduce brain response to visual food cues in humans. We hypothesize that exendin-[9-39] will diminish the effect of a meal in suppressing subsequent food intake and in reducing activation to visual food cues in reward pathways. Determining the extent to which the experience of satiety arises from a decrease in the reward value of food is fundamentally important to understanding human feeding behavior. In addition, this promising line of research is directly relevant to some of the most pressing public health issues of our time: obesity and overnutrition. We hope that investigating mechanisms affecting our perception of satiety at the most basic level will eventually result in novel behavioral or pharmacologic strategies for obesity prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18-29 years of age
2. BMI between 18.5-24.9 kg/m2
3. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Chronic health conditions, including diabetes and kidney disease.
2. Current dieting for weight loss or restrained eating
3. History of obesity, eating disorders, or weight loss surgery
4. Random blood glucose >140
5. Pregnancy or use of oral contraceptives
6. Current smoker
7. Recreational drug use or alcohol use of > 1 drink per day for females, > 2 per day for males
8. Food allergy or intolerance to study foods.
9. Medications known to alter appetite (e.g., amphetamines, atypical antipsychotics) or gastric emptying (e.g., metoclopromide)
10. Contraindications to MRI, such as implanted metal or claustrophobia.
11. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Study 1 - Amount of food eaten at a lunch buffet | 1 year
Study 2 - BOLD response as measured by fMRI during viewing of food photographs | 1 year

SECONDARY OUTCOMES:
Study 1 - Patient-reported appetite and appeal ratings | 1 year
Study 2 - Amount of food eaten at a lunch buffet and self-reported appetite ratings | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ellen A Schur, M.D., M.S., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Melhorn SJ, Tyagi V, Smeraglio A, Roth CL, Schur EA. Initial evidence that GLP-1 receptor blockade fails to suppress postprandial satiety or promote food intake in humans. Appetite. 2014 Nov;82:85-90. doi: 10.1016/j.appet.2014.07.009. Epub 2014 Jul 15. PMID 25049134